CLINICAL TRIAL: NCT05367388
Title: An Open-Label, Multi-Center, Randomized, 2-Way Crossover Study to Assess the Bioequivalence of APL-101 Capsule vs PLB-1001 Capsule in Healthy Chinese and Caucasian Subjects
Brief Title: A Study Comparing Two Different Capsules, APL-101 and PLB-1001 Capsules, in Healthy Chinese and Caucasian Participants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Apollomics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: APL-101-03
Record Dates: First submitted 2022-05-03; First posted 2022-05-10 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Bioequivalence
Keywords: Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: The treatment sequence will be determined using a 2×2 crossover design. This study includes an adaptive design feature of variable sample size.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence A/P (Experimental): Subject will receive a single oral dose (200mg) of Treatment A on Day 1, followed by a 7-day washout period. On Day 8, the subject will begin the second treatment period by receiving a single oral dose (200 mg) of Treatment P.
  Interventions: Drug: APL-101; Drug: PLB-1001
- Treatment Sequence P/A (Experimental): Subject will receive a single oral dose (200mg) of Treatment P on Day 1, followed by a 7-day washout period. On Day 8, the subject will begin the second treatment period by receiving a single oral dose (200 mg) of Treatment A.
  Interventions: Drug: APL-101; Drug: PLB-1001

INTERVENTIONS:
Drug: APL-101 — APL-101 (Vebreltinib) is an orally available small molecule, which is a tyrosine kinase inhibitor (TKI) for the mesenchymal epithelial transition protein tyrosine kinase receptor (c-Met) with high selectivity and potency.
  The treatments to be administered in this study include:
  • Treatment A (reference): Two 100 mg APL-101 (Vebreltinib) capsules (200 mg dose), manufactured for Apollomics, Inc.
  Other Names: Bozitinib; Vebreltinib
Drug: PLB-1001 — PLB-1001 (Bozitinib) is a chemical drug category 1.1 innovative drug. It is a highly effective and highly selective c-Met tyrosine kinase inhibitor.
  The treatments to be administered in this study include:
  • Treatment P (test): Two 100 mg PLB-1001 (Bozitinib) capsules (200 mg dose), manufactured for Beijing Pearl Biotechnology Co., Ltd.
  Other Names: Bozitinib

SUMMARY:
This is a Phase 1, open-label, multi-center, randomized, 2-period, adaptive design, crossover study to assess the bioequivalence of APL-101 (Vebreltinib) capsules and PLB-1001 (Bozitinib) capsules.

The treatments to be administered orally in this study include:

* Treatment A (reference): Two 100 mg APL-101 (Vebreltinib) capsules (200 mg dose), manufactured for Apollomics, Inc
* Treatment P (test): Two 100 mg PLB-1001 (Bozitinib) capsules (200 mg dose), manufactured for Beijing Pearl Biotechnology Co., Ltd.

APL-101 capsules (Treatment A) and PLB-1001 capsules (Treatment P) are similar drug products.

DETAILED DESCRIPTION:
Up to 48 healthy male subjects (approximately 16 Chinese and approximately 32 Caucasians) will be enrolled in the study in at least 2 sequential cohorts and randomly assigned to 1 of 2 treatment sequences. The treatment sequence will be determined using a 2×2 crossover design. This study includes an adaptive design feature of variable sample size. Data from the first 16 subjects will be used to determine the intra-subject variability to ensure a sufficient total sample size to achieve study objectives. If needed, up to 72 subjects will be enrolled.

ELIGIBILITY:
Major Inclusion Criteria:

* Must be Chinese (1st generation or 2nd generation Chinese with both Chinese parents), or Caucasian.
* Body mass index between 18.0 and 30.0 kg/m2, inclusive.
* In good health, determined by no clinically significant findings from medical history, physical examination, 12 lead ECG, vital sign measurements, and clinical laboratory evaluations at screening and at check-in as assessed by the Investigator (or designee). Screening clinical laboratory evaluations may be repeated once at the discretion of the Investigator.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 1.5 × the upper limit of normal (ULN), total bilirubin ≤ 1.5 × ULN at screening and check-in. Subjects with ALT or AST >1.0 × ULN combined with total bilirubin >1.0 × ULN are excluded.
* QT interval corrected for heart rate using Fridericia's method (QTcF) ≤ 450 msec confirmed by calculating the mean of the triplicate measurements within 4 weeks prior to Day 1.
* Systolic blood pressure between 100 and 140 mmHg or diastolic blood pressure between 50 and 90 mmHg, confirmed by calculating the mean of the triplicate measurements within 4 weeks prior to Day 1.

Major Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator.
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator.
* Have positive Coronavirus Disease 2019 (COVID-19) test at screening and/or at check-in, have clinical signs or symptoms of COVID-19 as determined by the Investigator, or have ongoing significant complication(s) from prior COVID-19 infection.
* Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant derived preparations within 14 days prior to check in, unless deemed acceptable by the Investigator.
* Have previously completed or withdrawn from this study or any other study investigating APL 101 or similar drug product, and/or have previously received APL 101 or similar drug product.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | Day 1 to Day 14
  Area under the curve (AUC) from time zero to infinity (AUC0-∞) and from time zero to the last quantifiable concentration (AUC0-last)
Maximum observed plasma concentration | Day 1 to Day 14
  Maximum observed plasma concentration (Cmax) after dosing of both treatments

SECONDARY OUTCOMES:
Time to the maximum observed plasma concentration | Day 1 to Day 14
  Time to the maximum observed plasma concentration (tmax)
Number of adverse events observed | Day 1 to Day 20-22
  Number of incidences of adverse events observed with respect to severity and relatedness to study treatment.
Apparent plasma terminal elimination half-life | Day 1 to Day 14
  Apparent plasma terminal elimination half-life (t1/2) after dosing of both treatments

CONTACTS AND LOCATIONS:
Overall Officials: Marietta Franco, MS, Study Director — Apollomics Inc.
Locations (1):
- New Zealand Clinical Research, Auckland, New Zealand